CLINICAL TRIAL: NCT01841905
Title: Detection of Disease-Related Changes in Pre-Symptomatic Alzheimer's Disease
Acronym: Scope
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Rhode Island Hospital (Other)
Collaborators: Pfizer (Industry); Heidelberg Engineering, Inc. (Unknown); Neurotrack (Unknown); Optovue (Industry); Avid Pharmaceuticals (Unknown)
Responsible Party: Sponsor
Other Study IDs: 900,421-477
Record Dates: First submitted 2013-04-24; First posted 2013-04-29 (Estimated); Last update posted 2016-01-20 (Estimated); Status verified 2016-01

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's Disease; Family History; Memory Concerns
MeSH Terms: conditions — Alzheimer Disease | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Observational Study: Pre-Symptomatic Alzheimers' Disease
  Interventions: Other: Observational Study

INTERVENTIONS:
Other: Observational Study — Observational Study

SUMMARY:
The investigators are conducting a study to try to improve our ability to identify older adults who are at high-risk for progression to Alzheimer's disease, several years before they have symptoms that might reduce their quality of life. The investigators believe they can increase the sensitivity of tests of memory and problem solving, by using a very small dose of a medication (scopolamine) that reduces the activity of the principal chemical system in the brain that is changing in the earliest stages of Alzheimer's disease. By pairing this "micro-dose" drug challenge (that is administered with a tiny needle placed just under the surface of the skin on the forearm), with our tests of memory and thinking, it is believed that the investigators can create a "stress test" that is very similar in concept to the use of the exercise treadmill to make the results of a heart EKG more sensitive to detect early disease, as a cardiac stress test for heart disease. The investigators want to create a similar stress test for Alzheimer's disease (AD).

DETAILED DESCRIPTION:
We will take pictures of subjects' brains using PET imaging, in healthy older adults (ages 55 to 80 years) who have both a family history of AD, and who have concerns about changes in their memory (but no clinical symptoms of AD), to see how much of a protein - that is related to AD -is in their brains. When all subjects come to the hospital for PET imaging, we will review the entire study plan with them, the risks and benefits of participation, and we will obtain written informed consent at that time. Our goal is to compare performance on our new stress test to these PET imaging results. Once the PET imaging is done, we will have each subject come to our clinical research unit for a day-long baseline visit. In the morning we will give the tests of memory and thinking, and then we will administer the injection of scopolamine at a very low dose. We will then continue to examine the subjects, and to give the memory and thinking tests at 1, 3, 5, 7, and 8 hours post-dosing. Once they have fully-recovered from all effects of the medication, they will be allowed to go home that day. We will then see all subjects again, for much shorter visits to complete the cognitive tests, at both 9 and 18 months after their initial study visit. We will follow all subjects for 18 months to see which of them show very mild but measurable changes on the memory and thinking tests, as we predict that these will be the same persons who also had stronger results on our stress test at the first study visit.

At all three study visits to our clinical research unit, we will obtain measurements using an imaging device that uses infrared and blue light to take picture of the eye and retina. Our secondary goal in this study to search for evidence of the same protein, in the retina, that builds up and is seen with PET imaging of the brain in persons who are at high risk for AD. Finally, we are also collecting a small sample of saliva, at the first visit to our unit, in order to see which subjects have a genetic risk for the disease, as this genetic risk may affect how we interpret the results of our new "cognitive stress test".

In this study, a small dose of an already approved medication (used to treat seasickness) will be used to temporarily, and safely, mimic signs of very early disease during just the first day of testing. This is a methodological study to determine if tests that measure how you think can predict the risk of dementia as we age.

ELIGIBILITY:
Inclusion Criteria:

* Individuals between the ages of 55 and 80 years old (inclusive).
* MMSE total score > 27
* Two risk factors for AD:
* Subjective memory complaints.
* A positive (suspected) first-degree family history for the disease.
* Permitted medications stable for at least 1 month prior to screening.
* Subjects may take stable doses of antidepressants lacking significant anticholinergic side effects (do not have a history of major depression within the past year).
* Estrogen replacement therapy.
* Adequate visual and auditory acuity to allow neuropsychological testing.
* Good general health or without any clinically significant abnormalities .
* Vitamin supplements (including Vitamin E) will be acceptable.
* Subjects must be willing and able to provide written informed consent.

Exclusion Criteria:

* History of major traumatic brain injury, other known neurologic disease or insult
* Mini Mental State Examination (MMSE)total score < 27
* Regular (daily) use of narcotics or antipsychotic medications
* Poorly-controlled major depression or another Axis I psychiatric disorder as described in DSM-IV within the past year.
* Psychotic features, agitation or behavioral problems, within the last 3 months.
* History of alcohol or substance abuse or dependence within the past 2 years (DSM IV criteria).
* History of schizophrenia (DSM IV criteria).
* Any significant systemic illness or unstable medical condition which could lead to difficulty complying with the protocol including:
* History of systemic cancer within the past 5 years (non-metastatic skin cancers are acceptable).
* History of myocardial infarction in the past year or unstable or severe cardiovascular disease including angina or Congestive Heart Failure (CHF) with symptoms at rest.
* Clinically significant obstructive pulmonary disease or asthma.
* Clinically significant and unstable gastrointestinal disorder within two years.
* Insulin-requiring diabetes or uncontrolled diabetes mellitus.
* Uncontrolled hypertension (systolic BP > 170 or diastolic BP > 100).
* History of clinically significant liver disease, coagulopathy, or vitamin K deficiency within the past 2 years.
* History of symptoms of narrow-angle glaucoma.
* Clinically significant obstructive uropathy
* Use of centrally active beta-blockers, narcotics, methyldopa and clonidine within 4 weeks prior to screening.
* Use of anti-Parkinsonian medications (e.g., Sinemet, amantadine, bromocriptine, pergolide and selegiline) within 2 months prior to screening.
* Use of neuroleptics or narcotic analgesics within 4 weeks prior to screening.
* Use of long-acting benzodiazepines or barbiturates within 4 weeks prior to screen.
* Use of short-acting anxiolytics or sedative-hypnotics more frequently than 2 times per week within 4 weeks prior to screening (note: sedative agents should not be used within 72 hours of the baseline and follow-up visits.
* Initiation or change in dose of an antidepressant lacking significant cholinergic side effects within the 4 weeks prior to screening (use of stable doses of antidepressants for at least 4 weeks prior to screening is acceptable)
* Use of systemic corticosteroids within 3 months prior to screening.
* Medications with significant cholinergic or anticholinergic side effects within 4 weeks prior to screening.
* Use of anti-convulsants within 2 months prior to screening.
* Use of warfarin (Coumadin) within 4 weeks prior to screening.
* Any prior use of any FDA approved medications for the treatment of Alzheimer's disease (e.g., tacrine, donepezil, or other newly approved medications).
* Use of any investigational drugs within 30 days or 5 half-lives, whichever is longer, prior to screening.
* Subjects who, in the investigator's opinion, will not comply with study procedures.
* Known hypersensitivity to F-18, tropicamide, and/or scopolamine or agents of this class of drugs.

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals between the ages of 55 and 80 years old, and who have two risk factors for AD (subjective memory complaints as ascertained on a standardized questionnaire and a positive family history for the disease).
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2013-07; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Groton Maze Learning Test | 18 Months
  Total number of correct moves over 5 trials on the Groton Maze Learning Test at 3 hours

SECONDARY OUTCOMES:
Groton Maze Learning Test | 18 Months
  Mean number of correct moves per second on the Groton Maze Learning Test at 3 hours
CogState One-Back Learning (OBK) Task | 18 Months
  Overall performance across study visits.
12-Item International Shopping List Test - Immediate and Delayed Recall (CogState) | 18 Months
  Overall performance across study visits.
Rentz Face-Name Association Test | 18 Months
  Overall performance across study visits.
Stark Pattern Separation Test | 18 Months
  Overall performance across study visits.
Minnesota Cognitive Acuity Scale (MCAS) | Pre-baseline
  Screening acuity.
Saliva Sample for DNA Analyses (ApoE and BDNF genotyping) | Baseline
  Mutation status.
Non-invasive imaging of macula, retinal function and visual fields | 18 Months
  Change over time.
CogState Once-Card learning (OCL) Task | 18 Months
  Overall performance across study visits.
Amyloid and Alzheimer's Psycho-educational Session | 9 and 18 month study visits
  An informational exercise to provide further information about amyloid PET imaging and to determine the impact of this disclosure of study participants.
Tokyo Subway Navigation | 9 month follow-up visit
  A functional activity of daily living where study participants are given pre-determined destinations / conditions and asked to map the route. Main outcome measure for this assessment is time taken to solve the problem.
MAC-Q | Pre-screen, Baseline, 9 & 18 month follow-up
  A six-item scale measuring age-related memory decline. An overall index of cognitive decline is calculated by summing scores for all six items with double weighting for item #6. Higher scores indicate greater decline in memory.

CONTACTS AND LOCATIONS:
Overall Officials: Peter J. Snyder, Ph.D., Principal Investigator — Sr. Vice President & Chief Research Officer, Lifespan
Locations (1):
- Lifespan, Providence, Rhode Island, United States